CLINICAL TRIAL: NCT01320332
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled Study to Assess the Pharmacokinetics, Safety, and Tolerability of ASP3291 Following a Single Oral Dose in Subjects With Ulcerative Colitis
Brief Title: A Study of a Single Dose of ASP3291 in Subjects With Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telsar Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3291-CL-0003
Record Dates: First submitted 2011-03-15; First posted 2011-03-22 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; ASP3291
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP3291 low dose (Experimental)
  Interventions: Drug: ASP3291
- ASP3291 high dose (Experimental)
  Interventions: Drug: ASP3291
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP3291 — Oral tablets
  Arms: ASP3291 high dose; ASP3291 low dose
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) and to assess safety and tolerability of a single dose of ASP3291 in subjects with ulcerative colitis.

DETAILED DESCRIPTION:
After an 11-day screening period, subjects check into a clinic, are dosed on Day 1 and stay in the clinic for 4 days to monitor pharmacokinetic and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a previously documented diagnosis of ulcerative colitis (UC) with endoscopy and histology consistent with diagnosis
* If female, the subject is at least 2 years postmenopausal or is surgically sterile per documentation provided by a third party medical professional or the subject agrees to use 2 highly effective methods of birth control during the study and is not pregnant or lactating
* Subject is willing and able to comply with the study requirements
* Subject has a body mass index (BMI) of <32 kg/m2
* Subject has ulcerative colitis requiring treatment with 5-aminosalicylic acid (5-ASA)

Exclusion Criteria:

* Subject has undergone previous resective colonic surgery
* Subject has previously diagnosed Crohn's Disease based on medical history
* Subject has an extension of disease limited to ulcerative proctitis
* Subject has active peptic ulcer disease based on medical history
* Subject is currently being treated with any prescription medication except the following: A stable dose of 5-aminosalicylic acid (5-ASA) for at least 2 weeks, oral contraceptives or hormone replacement therapy (HRT)
* Subject has a history of human immunodeficiency virus (HIV)
* Subject has a history of severe allergic or anaphylactic reactions
* Subject has a history of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment through analysis of blood, fecal and urine samples | Up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (3):
- United States (3):
  - Advanced Clinical Research Institute, Anaheim, California
  - SNBL Clinical Pharmacology Center, Baltimore, Maryland
  - Clinical Trials of Texas, Inc., San Antonio, Texas